CLINICAL TRIAL: NCT05212220
Title: Low-intensity Ecological Momentary Assessment (EMA) for Smoking Cessation Intervention and Tobacco Control Policy Evaluation: a Randomized Controlled Trial Nested Within an EMA-based Observational Study
Brief Title: Effectiveness of Ecological Momentary Assessment Based Smoking Cessation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05190077
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2023-05

CONDITIONS: Smoking Cessation
Keywords: Ecological Momentary Assessment; Intervention; Smoking Cessation; Acceptance and commitment therapy; Unassisted quitting; Tobacco control policy
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will first receive 5 times EMA per day for one week. The EMA will document participants smoking behaviors, smoking cues, smoking cravings, etc. The intervention group will receive 15-30 minutes of a nurse-led phone call, and 10-week instant messaging after completing the one-week EMA documentation.
  Interventions: Behavioral: EMA-based intervention
- Control (No Intervention): The control group will first receive 5 times EMA per day for one week. The EMA will document participants smoking behaviors, smoking cues, smoking cravings, etc. No intervention will be provided to the control group after completing the one-week EMA documentation.

INTERVENTIONS:
Behavioral: EMA-based intervention — A personal quit plan includes (1) self-help techniques on handling craving; (2) suggestions to avoid the reported pro-smoking cues; (3) whether to quit progressively or abruptly; (4) referral for existing smoking cessation service; and (5) instruction of using over-the-counter (OTC) nicotine replacement therapy (NRT), if OTC-NRT is preferred by the participant will be designed and give to the participants via a nurse-led phone call.
  Arms: Intervention
Behavioral: EMA-based intervention — Participants will receive 10-week tailored quitting reminder instant messages via WhatsApp and voluntarily discuss their quit plan with the research staff.
  Arms: Intervention

SUMMARY:
The EMA-based intervention in this proposal is aimed to motivate the majority of smokers who do not prefer to use traditional cessation aids for quitting and help them quit smoking. The smartphone application (app) and the EMA-based phone reminders at low cost and short intervention time make this approach attractive for the majority of smokers. Identification of accurate and specific pro-smoking cues in the real-word and real-time environmental cues via the app will provide valuable information to guide new tobacco control policies.

DETAILED DESCRIPTION:
Study design:

The proposed study comprises a 2-arm (allocation ratio 1:1) RCT to assess the efficacy of the EMA-based smoking cessation intervention and the EMA-based observational study. Throughout the 7-day participation, all recruited participants will complete an EoD survey and 4 time-based system-triggered EMA each day. The surveys will be prompted by a smartphone application (app) installed in their own mobile phones. The prompting time will be personalized and pre-scheduled by the participants. The information collected in the app will be used to develop an EMA-based intervention including a quit plan and 10-week quitting reminders and for an EMA-based observational study. I will randomly allocate half of the participants (intervention group) to receive the EMA-based intervention. All participants will then be contacted for a follow-up at 3- and 6-month.

Subjects:

This proposed study aims to recruit daily tobacco users, regardless of intention to quit.The inclusion criteria are: (1) daily consumption of tobacco products (including traditional cigarettes, electronic cigarettes, and heated tobacco products) in the past week; (2) age ≥18 years; (3) owning a mobile smartphone with internet access; (4) staying in Hong Kong during the 1-week EMA study period; and (5) able to read and write Chinese. Participants' smoking status will be confirmed by measuring exhaled carbon monoxide to be 4ppm or above, or saliva cotinine to be 30ng/ml or above. Because the proposed study aims to promote smoking cessation in smokers who do not plan to use smoking cessation aids, we will exclude smokers who (1) plan to use smoking cessation services or medication in the coming month or (2) using smoking cessation services, or using nicotine replacement therapy in the past 7 days. Smokers who reported having mental illnesses and female smokers who are pregnant are also excluded as they need more specific smoking cessation intervention.

Recruitment procedures:

Recruitment will be conducted both offline and online. In the outdoor recruitment, the recruitment staff first approach and distribute souvenirs (e.g., a tissue pack) to the smokers at outdoor smoking hotspots. If the smoker is willing to accept souvenirs and talk to the recruitment staff, the staff will ask further questions related to eligibility. Eligible participants will: (1) be given more detail about this project, (2) be invited to provide written consent, (3) be assisted in installing EMA app on their mobile phone and setting EMA schedule, (4) complete baseline questionnaire by paper form or Qualtrics. Due to the time-limited at outdoor recruitment, participants can complete baseline questionnaire after the recruitment session.

Research assistants will also send mass emails or advertisements through social media (e.g., Facebook, Instagram). Potential participants who are interested in this project can scan the QR code on the advertisement and complete the online application form (using Qualtrics). Our recruitment staff makes appointments with the potential participants to complete the recruitment procedures.

Ecological momentary assessment:

An EMA app will be developed to document all smoking cues and smoking-related behaviors. After installing the EMA app on participants' smartphones, participants need to input the five last digit numbers of their telephone number as an identifier and select the date they would like to start the EMA survey. Participants need to complete 5 time-based EMA surveys per day for 7 consecutive days, each EMA survey with an interval of three hours.

The EMA questions on smoking cues cover 4 domains: emotional, social, pattern, and withdrawal cues. Smoking-related behaviors include (1) smoking tobacco (traditional cigarettes, heated tobacco products, and electronic cigarettes) during the past 3 hours, (2) nicotine craving during the past 3 hours and type of craving (physical, psychological or social craving), (3) purchasing tobacco products during the past 3 hours. Whether the smoking-related behaviors have been due to the exposure to the pro-smoking cues will also be asked. Sleep quality will be asked by (1) did you experience insomnia problem (difficulty falling asleep, difficulty staying asleep, problems waking up too early) for last night (none, mild, moderate, severe, very severe), (2) how satisfied are you with your last night sleep pattern (score range from 0 very satisfied to 4 very dissatisfied) in first EMA for each day. 'Time to consume the first cigarette after waking' will be asked at the second EMA. Tobacco control policy, including health warnings on their tobacco pack; POS tobacco displays; smoking hotspots, and daily tobacco consumption, will be asked at the last EMA for each day.

Intervention:

Based on the EMA of each participant, a trained research nurse will review their (1) nicotine dependence; (2) intensity and frequency of reported cravings; and (3) the impact of exposure to pro-smoking cues on smoking behaviors. A personalized quit plan will be developed based on tailored suggestions from the US clinical practice guideline for smoking cessation, Smoking Cessation Information Kit (published by Department of Health), the theory of Health Action Process Approach, and the self-determination theory. Our recent studies showed that interventions based on these theories are effective. Half of the randomly selected participants (intervention group) will receive this quit plan via a nurse-led phone call, email, and WhatsApp. The nurse will then design a quit plan including (1) self-help techniques on handling craving; (2) suggestions to avoid the reported pro-smoking cues; (3) whether to quit progressively or abruptly; (4) referral for existing smoking cessation service; and (5) instruction of using over-the-counter (OTC) nicotine replacement therapy (NRT), if OTC-NRT is preferred by the participant. Participants will then receive tailored quitting reminders via WhatsApp and voluntarily discuss their quit plan with the nurse in the subsequent 10 weeks.

Randomization, blinding, and allocation concealment:

The research staff will randomly assign participants on an individual level to intervention and control group using a 1:1 allocation ratio by sequentially numbered, opaque sealed envelope method. The principle will generate a list of random numbers using the random function of Excel. Then prepare about 450 identical, opaque, sealed, A5-sized envelopes, with a unique 3-digit serial number on the cover of each envelope as an identifier, and put the allocation code into the envelopes. All recruitment staff and participants will be concealed to the group allocation at recruitment. After a participant consents to the trial, the research staff will retrieve his/her information and open 1 envelope to allocate the recruited participant according to the card inside.

Participants and research staff of intervention delivery will not be blinded to the intervention because the intervention is behaviors. However, assessors of the follow-up and the research investigators will not be involved in the recruitment and intervention delivery and will be blinded to the group allocation (i.e. single-blinded design).

Follow-up All participants will be followed up via telephone by an allocation-blinded interviewer at 3- and 6-month after consenting to participation. Only the participants who report abstinence in the past 7 days will be invited to measure their exhaled CO with a Smokerlyzer and/or saliva cotinine level with a Cotinniene Saliva Test Device at their residence, workplace, or nearby, according to their preference.

Sample size:

To date, there was no previous RCT that used EMA results to guide personalized nurse-led telephone counseling and instant messaging for smoking cessation. The effect size for personalized counseling and instant messaging was derived from a network meta-analysis. The sample size was calculated based on an anticipated intervention effect of an OR of 2.92 from the meta-analysis of tailored text messaging combined with counseling for smoking cessation. One of our previous RCTs showed that the prevalence of 3-month biochemically validated tobacco abstinence among Hong Kong smokers was 4% in the group receiving brief advice. To detect a significant difference of quit rate between two groups with a power of 80% (to reduce type II error) at 5% significant level (type I error), a total of 444 participants (allocation ratio 1:1; 222 vs 222) is needed.

Data analysis:

The primary analysis will examine the effect of EMA-based intervention on biochemically validated abstinence at 3-month and the difference in the IBC-S score between the two groups. Intention-to-treat approach will be used to include all consented participants in the analysis and assume non-respondents at the 3-month follow-up as smokers and no change on the IBC-S score. A generalized estimating equation (GEE) analysis with exchangeable structure for the correlation matrix will be used for biochemically validated abstinence after adjusting unbalance baseline demographics and other variables that have been reported to be associated with smoking cessation. We will use linear regression adjusted for imbalance socio-demographics assessed at baseline to compare the score of IBC-S between intervention and control groups. Multiple imputation will be used to deal with missing values for baseline socio-demographics. All secondary and ancillary outcomes will be analyzed with either GEE (binary outcomes) or linear mixed models (continuous outcomes). Subgroup analysis of comparing the primary and secondary outcomes between intervention group participants who received both nurse-led phone calls plus instant messaging and instant messaging only will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Daily consumption of tobacco products (including traditional cigarettes, electronic cigarettes, and heated tobacco products) in the past week;
2. Age ≥18 years;
3. Owning a mobile smartphone with internet access;
4. Staying in Hong Kong during the 1-week EMA study period;
5. Able to read and write Chinese
6. Exhaled carbon monoxide will be measured and required to be 4ppm or above, or saliva cotinine to be 30ng/ml or above

Exclusion Criteria:

1. Plan to use smoking cessation services or medication in the coming month
2. Using smoking cessation services, or using nicotine replacement therapy in the past 7 days
3. Having mental illnesses
4. Female smokers who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Incremental Behavior Change Towards Smoking Cessation (IBC-S) at 3-month follow-up | 3-month follow-up
  Behavioral progression towards smoking cessation will be detected by 15-item Incremental Behavior Change towards Smoking Cessation. 15-item Incremental Behavior Change towards Smoking Cessation contains two parts: behavioral and cognitive changes. Item 1 to Item 12 are binary questions on a scale of 0 to 1 (0, no; 1, yes) to evaluate the behavioral changes. Cognitive changes are measured by item 13 to 15 on a scale of 0 to 4 (0, not at all; 4 always). Higher score means a better outcome.
Prevalence of biochemical validated abstinence at 3-month follow-up | 3-month follow-up
  Tobacco abstinence in the past 7 days, which is validated using an exhaled carbon monoxide level of< 4 ppm, and a saliva cotinine level of < 30 ng/ml.
  Noted:
  1. Suppose participants refuse to have a face-to-face exhaled carbon monoxide test due to the pandemic of COVID-19 in Hong Kong. In that case, the outcome will be validated by a cotinine saliva test device only.
  2. If participants use NRT, the outcome will be validated by exhaled carbon monoxide only.

SECONDARY OUTCOMES:
Prevalence of biochemical validated abstinence at 6-month follow-up | 6-month follow-up
  Tobacco abstinence in the past 7 days, which is validated using an exhaled carbon monoxide level of< 4 ppm, and a saliva cotinine level of < 30 ng/ml.
  Noted:
  1. Suppose participants refuse to have a face-to-face exhaled carbon monoxide test due to the pandemic of COVID-19 in Hong Kong. In that case, the outcome will be validated by a cotinine saliva test device only.
  2. If participants use NRT, the outcome will be validated by exhaled carbon monoxide only.
Prevalence of self-reported 7-day abstinence at 3-month follow-up | 3-month follow-up
  Self-reported 7-day abstinence at 3-month follow-up
Prevalence of self-reported 7-day abstinence at 6-month follow-up | 6-month follow-up
  Self-reported 7-day abstinence at 6-month follow-up
Self-reported use of smoking cessation service or medication from baseline at 3-month follow-up | 3-month follow-up
  Use of smoking cessation service or medication from baseline at 3-month follow-up

OTHER OUTCOMES:
Self-report quit attempts at 3-month follow-up | 3-month follow-up
  Number of quit attempts from baseline at 3-month follow-up
Self-efficacy to quit smoking at 3-month follow-up | 3-month follow-up
  Self-efficacy will be evaluated according to the importance of quitting on a scale of 0 to 10 (0, least important; 10, most important), the difficulty of quitting on a scale of 0 to 10 (0, least difficult; 10, most difficult), and confidence in quitting on a scale of 0 to 10 (0, least confident; 10, most confident). For the scale of measuring quitting importance and confidence, higher scores mean a better outcome and for the scale of measuring difficulty, higher scores mean a worse outcome.
Self-report satisfaction toward instant messages at 3-month follow-up | 3-month follow-up
  Defined by rating the satisfaction of instant messages on a scale of 0 to 4 (0, very dissatisfied; 4 very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years after the completion of the relevant publications.

REFERENCES:
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Result] Cheung YTD, Lam TH, Li WHC, Wang MP, Chan SSC. Feasibility, Efficacy, and Cost Analysis of Promoting Smoking Cessation at Outdoor Smoking "Hotspots": A Pre-Post Study. Nicotine Tob Res. 2018 Nov 15;20(12):1519-1524. doi: 10.1093/ntr/ntx147. PMID 28655173
- [Result] Chan SS, Wong DC, Cheung YT, Leung DY, Lau L, Lai V, Lam TH. A block randomized controlled trial of a brief smoking cessation counselling and advice through short message service on participants who joined the Quit to Win Contest in Hong Kong. Health Educ Res. 2015 Aug;30(4):609-21. doi: 10.1093/her/cyv023. Epub 2015 Jun 25. PMID 26116584
- [Result] Cheung YT, Wang MP, Li HC, Kwong A, Lai V, Chan SS, Lam TH. Effectiveness of a small cash incentive on abstinence and use of cessation aids for adult smokers: A randomized controlled trial. Addict Behav. 2017 Mar;66:17-25. doi: 10.1016/j.addbeh.2016.11.006. Epub 2016 Nov 10. PMID 27863323
- [Result] Hartmann-Boyce J, Livingstone-Banks J, Ordonez-Mena JM, Fanshawe TR, Lindson N, Freeman SC, Sutton AJ, Theodoulou A, Aveyard P. Behavioural interventions for smoking cessation: an overview and network meta-analysis. Cochrane Database Syst Rev. 2021 Jan 4;1(1):CD013229. doi: 10.1002/14651858.CD013229.pub2. PMID 33411338
- [Result] Hernandez-Lopez M, Luciano MC, Bricker JB, Roales-Nieto JG, Montesinos F. Acceptance and commitment therapy for smoking cessation: a preliminary study of its effectiveness in comparison with cognitive behavioral therapy. Psychol Addict Behav. 2009 Dec;23(4):723-30. doi: 10.1037/a0017632. PMID 20025380
- [Result] Wang MP, Luk TT, Wu Y, Li WH, Cheung DY, Kwong AC, Lai V, Chan SS, Lam TH. Chat-based instant messaging support integrated with brief interventions for smoking cessation: a community-based, pragmatic, cluster-randomised controlled trial. Lancet Digit Health. 2019 Aug;1(4):e183-e192. doi: 10.1016/S2589-7500(19)30082-2. Epub 2019 Jul 31. PMID 33323188
- [Result] Hoeppner BB, Hoeppner SS, Abroms LC. How do text-messaging smoking cessation interventions confer benefit? A multiple mediation analysis of Text2Quit. Addiction. 2017 Apr;112(4):673-682. doi: 10.1111/add.13685. Epub 2016 Dec 12. PMID 27943511
- [Result] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Result] Yu DS. Insomnia Severity Index: psychometric properties with Chinese community-dwelling older people. J Adv Nurs. 2010 Oct;66(10):2350-9. doi: 10.1111/j.1365-2648.2010.05394.x. Epub 2010 Aug 16. PMID 20722803
- [Result] Cropsey KL, Trent LR, Clark CB, Stevens EN, Lahti AC, Hendricks PS. How low should you go? Determining the optimal cutoff for exhaled carbon monoxide to confirm smoking abstinence when using cotinine as reference. Nicotine Tob Res. 2014 Oct;16(10):1348-55. doi: 10.1093/ntr/ntu085. Epub 2014 Jun 2. PMID 24891552
- [Result] Cooke F, Bullen C, Whittaker R, McRobbie H, Chen MH, Walker N. Diagnostic accuracy of NicAlert cotinine test strips in saliva for verifying smoking status. Nicotine Tob Res. 2008 Apr;10(4):607-12. doi: 10.1080/14622200801978680. PMID 18418783
- [Result] Flocke SA, Step MM, Lawson PJ, Smith S, Zyzanski SJ. Development of a Measure of Incremental Behavior Change Toward Smoking Cessation. Nicotine Tob Res. 2017 Dec 13;20(1):73-80. doi: 10.1093/ntr/ntw217. PMID 27613910
- [Result] Gilbert H, Sutton S, Morris R, Petersen I, Galton S, Wu Q, Parrott S, Nazareth I. Effectiveness of personalised risk information and taster sessions to increase the uptake of smoking cessation services (Start2quit): a randomised controlled trial. Lancet. 2017 Feb 25;389(10071):823-833. doi: 10.1016/S0140-6736(16)32379-0. Epub 2017 Jan 25. PMID 28129989
- [Result] Casagrande JT, Pike MC. An improved approximate formula for calculating sample sizes for comparing two binomial distributions. Biometrics. 1978 Sep;34(3):483-6. No abstract available. PMID 719125
- [Result] Shiffman S. Conceptualizing analyses of ecological momentary assessment data. Nicotine Tob Res. 2014 May;16 Suppl 2(Suppl 2):S76-87. doi: 10.1093/ntr/ntt195. Epub 2013 Dec 9. PMID 24323571
- [Derived] Cheung YTD, Zhang MJ, Luk TT, Ho SY, Lam TH, Wang MP. Telephone Counseling and Messaging Guided by Mobile Profiling of Tobacco Users for Smoking Cessation: A Randomized Clinical Trial. JAMA Netw Open. 2025 Mar 3;8(3):e250764. doi: 10.1001/jamanetworkopen.2025.0764. PMID 40085082
- [Derived] Zhang MJ, He WJA, Luk TT, Wang MP, Chan SSC, Cheung YTD. Effectiveness of personalized smoking cessation intervention based on ecological momentary assessment for smokers who prefer unaided quitting: protocol for a randomized controlled trial. Front Public Health. 2023 Jul 31;11:1147096. doi: 10.3389/fpubh.2023.1147096. eCollection 2023. PMID 37583881